CLINICAL TRIAL: NCT05894057
Title: Observational Study to Understand Acceptability of Various Available Midazolam Formulations (Syrup, Rectal Suppository, Oro-dispersible Tablet) in Clinical Practice
Brief Title: Acceptability of Various Available Midazolam Formulations (Syrup, Rectal Suppository, Oro-dispersible Minitablet) in Clinical Practice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00302; ks22Pfister2
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Medication Palatability
Keywords: midazolam; midazolam oral syrup; midazolam rectal suppository; midazolam oro- dispersible mini-tablet; drug-adherence in pediatrics; pediatric sedation management; anxiolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (reference: midazolam oral syrup or rectal suppository formulations): Oral syrup or rectal suppository formulation of midazolam prescribed in the Anesthesiology Unit or Emergency Unit of UKBB as current reference formulations in clinical routine.
  Interventions: Other: Data collection on acceptability of midazolam administration by 2- to 10-year-old pediatric patients at UKBB
- Group 2 (alternative: midazolam oro- dispersible mini-tablet (OMDT) formulation): ODMT formulation of midazolam prescribed in the Anesthesiology or Emergency Unit at UKBB as a recently introduced alternative formulation in clinical routine.
  Interventions: Other: Data collection on acceptability of midazolam administration by 2- to 10-year-old pediatric patients at UKBB

INTERVENTIONS:
Other: Data collection on acceptability of midazolam administration by 2- to 10-year-old pediatric patients at UKBB — On the day of entry to the Anesthesiology Unit for an elective surgery, or before an intervention at the Emergency Unit, all children, irrespective of their participation to the present study, will receive standard midazolam dose of 0.3-0.5 mg/kg as prescribed by the treating clinician at UKBB in line with clinical practice (as oral syrup, rectal suppository or ODMT). The children's spontaneous reactions after intake of midazolam (e.g., positive comments, spitting out of medication, crying) will be observed and recorded by the research staff. Children who are able to understand the Hedonic Scale (FHS) will be questioned on how they liked the medication by pointing to the appropriate face of a Facial Hedonic Scale (FHS) at the time of midazolam intake.

SUMMARY:
This observational study aims to gain knowledge on how the different midazolam formulations (oral syrup, rectal suppository, ODMT) are accepted by 2- to 10-year-old pediatric inpatients and outpatients at the University Children's Hospital Basel (UKBB) in Switzerland. The present study will use non-invasive scoring to assess acceptability of the different midazolam formulations.

DETAILED DESCRIPTION:
At the University Children's Hospital Basel (UKBB) in Switzerland, ~ 2500 children are referred to the Pediatric Anesthesiology Unit per year receiving midazolam sedation before surgery. Further, ~2000 children are admitted to the Pediatric Emergency Unit for procedures requiring midazolam sedation per year. Medication palatability is a key element of treatment adherence and successful therapy outcome. In a previous cross-sectional acceptability study in 2- to 10-year-old pediatric patients at UKBB, it was demonstrated that an inorganic calcium carbonate/calcium phosphate carrier material as the main excipient in an oro- dispersible mini-tablet (ODMT) formulation is safe, palatable, and highly acceptable in children. To date, no data for acceptability in terms of palatability and anxiolysis in daily preoperative practice for midazolam oral syrup, rectal suppository or ODMT formulation is available. As such the goal of this observational study is to better understand acceptability of various midazolam formulations (oral syrup, rectal suppository, ODMT) in clinical practice in 2- to 10-year-old pediatric patients at UKBB. .

ELIGIBILITY:
Inclusion Criteria:

* Children from 2 years (meaning 2 years 0/12 months) to younger than 10 years (meaning 9 years 12/12 months) of age at the time of surgery
* Children scheduled for ambulatory or elective surgery or for procedures requiring anxiolysis at the UKBB
* Children qualifying as American Society of Anesthesiologists (ASA) 1 or ASA 2 patients
* Clinically indicated administration of midazolam oral syrup, rectal suppository or ODMT
* Parent or legal guardian has been informed about the study and has signed the Informed Consent Form

Exclusion Criteria:

* Children qualifying as ASA 3 and above patients
* Children arriving at the emergency ward in a critically ill condition which needs immediate intervention (i.e. American Thoracic Society (ATS) Score 1 and 2) and no tolerance for time delay due to informed consent.
* Difficulty in assessing palatability due to neurological impairments
* Hypersensitivity to midazolam, other benzodiazepines, or any formulation excipients
* Hypersensitivity to cherries (syrup)

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 2- to 10-year-old pediatric patients in the Pediatric Anesthesiology Unit and Pediatric Emergency Unit at the UKBB. Pediatric patients undergoing elective surgical or emergency procedures requiring anxiolysis with midazolam during clinical routine will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Children's acceptance after intake of midazolam rated by research staff | one time assessment at baseline
  4-point acceptability scale (from "child liked the medication" to "child did not like the medication") rated by research staff
Children's acceptance after intake of midazolam rated by the pediatric patients | one time assessment at baseline
  Children who are able to understand the Facial Hedonic Scale (FHS) will be questioned on how they liked the medication by pointing to the appropriate face of a Facial Hedonic Scale (FHS) at the time of midazolam intake. Each face will be associated to a number from a scale to 1 (very bad) to 6 (very good). The spontaneous reactions of the patient will be recorded to identify acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Beglinger, Dr. med., Principal Investigator — University of Basel Children's Hospital (UKBB)
Locations (1):
- University of Basel Children's Hospital (UKBB), Basel, Switzerland